CLINICAL TRIAL: NCT06237855
Title: Empowering Patients: A Randomized Controlled Trial (RCT) Investigating the Feasibility and Outcomes of Patient Self-Drain Removal After Ventral Hernia Repair
Brief Title: Investigating the Feasibility and Outcomes of Patient Self-Drain Removal After Ventral Hernia Repair
Acronym: SDR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the institution and no other investigator wants to continue the study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00100883
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-03

CONDITIONS: Ventral Hernia
Keywords: hernia repairs; drain removal; subcutaneous drains
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Comparison of control group (drain removal in clinic via provider) versus intervention group self-removing drain at home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Drain removal will occur during clinic visit by provider per standard of care procedure.
- Self-drain removal training (Experimental): Subjects will remove drain at home Training will consist of a detailed online video of a provider instructing how to remove the drain and practicing on a model created specifically to mimic the following actions during drain self-removal:
  * Tension required to remove the drain
  * Placing and taping gauze after suture and drain removal
  Interventions: Other: Self-drain removal

INTERVENTIONS:
Other: Self-drain removal — Subjects will be trained to self-remove drain at home following ventral hernia repair.
  Arms: Self-drain removal training

SUMMARY:
The goal of this randomized controlled trial is to teach patients to safely and effectively self-remove drains at home in adults (aged 18 and older) following a ventral hernia repair (VHR). Researchers will compare the group of subjects self-removing the drain at home to a control group of standard of care drain removal during a clinic visit by a provider to see if subjects are able to safely self-remove the drain at home.

DETAILED DESCRIPTION:
Annually, in the United States, it is estimated that 500,000 ventral hernia repairs (VHRs) are performed with a cost in excess of $3.2 billion. Drains are frequently used in an effort to prevent seroma formation. Seromas are defined as a buildup of bodily fluid in a potential space post-surgery, usually at the surgical site. Rate of seroma has been estimated to be between 9-11% following abdominal wall reconstruction (AWR). The timing of the removal is usually after discharge but before patient's scheduled postoperative visit, thus most patients must call and speak to a health provider and come in for an additional clinic visit specifically for drain removal. The goal of this study is to teach patients to safely and effectively self-remove drains at home. This will allow patients to forgo the cost associated with commuting to the clinic, the clinic cost associated with nursing time and scheduling, the clinic visit, physician or nurse time to remove the drain and possibly lost wages for the patient from time off work. It is important to note that self-drain removal will not compromise or deviate from typical patient follow up. Instead, this will eliminate an extra patient visit when inevitably the timing of drain removal does not align with the typical follow-up period. Additionally, this will allow providers to see additional patient consultations or perform other duties, as they will not have the time constraints associated with in-office drain removal. This study will show that patient self-drain removal benefits the patients, the providers, and healthcare system without compromising patient safety, satisfaction, and postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Undergoing elective ventral hernia repair (VHR).
* Sub-cutaneous drain placement.
* Anticipated Centers for Disease Control and Preventions (CDC) 1&2 wound class.

Exclusion Criteria:

* Patients who do not have access to the online training video.
* The surgeon does not believe the patient can self-remove the drain.
* Planned concomitant procedures.
* Current mesh infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Success rate of patients self-removing drains | 2 weeks post-operatively
  Percentage of patients that are able to safely self-remove drain at home.

SECONDARY OUTCOMES:
Wound complication rate | 30-days post-operatively.
  Comparison of the wound complication rate between the control and intervention groups. Wound complications will be defined as wound breakdown, wound cellulitis, hematoma, wound infection, and seroma requiring intervention. Each wound complication will be reported individually and as an aggregate wound complication overall rate.
Change in drain removal training survey scores from pre to post training | Hour 1
  Change in drain removal training survey scores from pre to post training. The same survey is given pre and post is training and is on a 5-point Likert scale survey with 1 representing "strongly disagree" and 5 representing "strongly agree". Higher scores indicate more confidence in the self-drain removing process.
Post-drain removal satisfaction survey scores | 30-days post-operatively
  Score on satisfaction survey following self-drain removal (intervention group only). Survey is on a 5-point Likert scale survey with 1 representing "strongly disagree" and 5 representing "strongly agree". Higher scores indicate greater satisfaction with at home self-drain removal.
Difference In Subject Costs | 30-days post-operatively
  Difference in cost associated with reduction in clinic visits.
Difference in Subject Amount of Time | 30-days post-operatively
  Difference in time associated with reduction in clinic visits and travel

CONTACTS AND LOCATIONS:
Overall Officials: Todd Heniford, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Laparoscopic & Advanced Surgery Program, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT06237855/ICF_000.pdf